CLINICAL TRIAL: NCT03130062
Title: Effectiveness of Resistance Exercise in Daily Motor Activity Index and Functional Fitness in Women With Primary Sjögren Syndrome: a Randomized Clinical Trial
Brief Title: Resistance Exercise in Woman With Primary Sjörgen Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Paulo Minali, Physical Education Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13041978
Record Dates: First submitted 2017-04-16; First posted 2017-04-26 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Primary Sjögren Syndrome
Keywords: Resistance Exercise; Functional Fitness; Actigraphy; Primary Sjögren Syndrome
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The division of the groups was obtained through randomization through a computer program. An opaque envelope containing the group allocation was given to the volunteer by the blind evaluator. After randomization, the sequential numbers were kept in opaque and closed envelopes and, as patients passed the initial evaluations, were allocated to one of the groups.
Who Masked: Outcomes Assessor
Masking Description: The collaborators who carried out these evaluations were unaware of the allocation of volunteers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Volunteers underwent a supervised resistance exercise program for 16 weeks. The subjects performed 10 exercises with 3 sets of 10 maximum repetitions in each. The training sessions were held twice a week.
  Interventions: Other: Exercise
- Control (No Intervention): Volunteers in this group were instructed not to perform systematic physical exercises for 16 weeks (the same period of the GEX group training program), and only the SSP medication treatment was maintained, and they were followed up during the study period.

INTERVENTIONS:
Other: Exercise — The following muscular clusters were exerted: latissimus dorsi, deltoid, pectoralis major , triceps brachialis, biceps brachialis, quadriceps, hamstring, thigh adductor muscles, thigh abductor muscles and gastrocnemius.
  Arms: Exercise

SUMMARY:
To analyze the effectiveness of 16-week resistance exercise in daily motor behavior and functional fitness in women with Primary Sjögren's Syndrome. The present study presents as hypothesis that a supervised resistance exercise program is effective and safe in improving the functional fitness and quality of life of patients with Primary Sjögren's Syndrome, making them more physically active, contributing positively to the capacity to perform daily life activities as household and / or professional tasks.

DETAILED DESCRIPTION:
Sjögren's syndrome (SS) is a systemic autoimmune inflammatory disease that affects the exocrine glands and less frequently the internal organs, presenting intense lymphoplasmacytic infiltration mainly in the epithelium of the involved tissues, leading to the destruction and loss of the secretory function. SS can manifest itself in isolation, without association with other diseases, in this situation it is called Primary Sjögren's Syndrome (PSS), being considered the second most common autoimmune rheumatic disease, prevalent in women (9: 1). The inflammatory process can affect any organ, resulting in a generally severe clinical condition, and may involve the musculoskeletal, pulmonary, gastrointestinal, hepatic, hematological, vascular, dermatological, renal and neurological systems, leading to an evident decline of the physical functions with decrease in aerobic capacity, muscular strength, joint mobility and static balance, as well as psychological and social deficit. Patients with PSS also present a marked physiological characteristic with a high level of fatigue. Thus, resistance exercise becomes a non-drug strategy, aiming to improve musculoskeletal fitness, allowing the execution of daily activities with more independence, autonomy and safety, while influencing the patient's functional fitness. The aim of the present study is to analyze the effectiveness of resistance exercise in daily motor behavior and functional fitness in women with Primary Sjögren's Syndrome. After the use of actigraphy for 15 days, equipment that measures the level of daily physical activity, and evaluation of functional fitness, volunteers underwent a supervised resistance exercise program for 16 weeks. The following muscular clusters were exerted: latissimus dorsi, deltoid, pectoralis major , triceps brachialis, biceps brachialis, quadriceps, hamstring, thigh adductor muscles, thigh abductor muscles and gastrocnemius. The subjects performed in each exercise 3 sets of 10 maximum repetitions. The training sessions were held twice a week.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of PSS - according to the criteria of the American-European Society for the classification of Primary Sjögren's Syndrome (Vitali et al., 2002);
* Female gender
* Aged above 18 years

Exclusion Criteria:

* Patients who had cognitive difficulties, with diagnosis of Secondary Sjögren's Syndrome,
* A regular physical exercise practitioner or who were practicing physical exercise regularly up to 2 months before the interview.
* Patients in clinical conditions that prevented the practice of physical exercise according to previous medical evaluation, such as decompensated diabetes mellitus, decompensated thyroid disease, severe cardiorespiratory diseases, etc. - Use of medications that interfere with physical aspects, especially in response to the sensation of fatigue.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in functional fitness | The subjects were assessed in 2 moments: before entering the resistance training program and after 16 weeks of intervention.
  The protocol consists of a sequence of 7 tests that aim to mimic the neuromotor and cardiorespiratory needs involved in the daily life activities. This battrey test was designed and validated to evaluate the elderly without a ceiling effect, ensuring that the physical aspect measured represents the maximum of the individual.
  The physiological components evaluated, based on the physical abilities performed in the daily activities are: upper and lower limb strength, aerobic capacity, upper and lower limb flexibility, as well as motor agility / dynamic balance. In addition, the authors added the body mass index (BMI), to estimate the body composition.
Change in daily motor activity index | The subjects were assessed for 15 consecutive days belonging to the habitual routine of the volunteers. It was used in 2 moments: before entering the resistance training program and after 16 weeks of intervention.
  To verify the daily movement index of the subjects we used a device called an actigraphy or actimeter.

SECONDARY OUTCOMES:
Quality of life estimate | The subjects were assessed in 2 moments: before entering the resistance training program and after 16 weeks of intervention.
  To evaluate the quality of life, the "Medical Outcomes Study SF-36", a generic questionnaire was translated and validated for the Brazilian population (Ciconelli, 1999). To evaluate, in a generic way, the quality of life. It is a multidimensional instrument composed of 36 items evaluating in 8 dimensions thus distributed: 10 items related to functional capacity; 4 physical appearance items; 2 items on pain; 5 items related to general health status; 4 items on vitality; 2 items with respect to social aspects; 3 items on emotional aspects; 5 items related to mental health and one more question of comparative evaluation between the current health conditions and that of a year ago.
Estimates of disease activity | The subjects were assessed in 2 moments: before entering the resistance training program and after 16 weeks of intervention.
  ESSDAI - Sjögren's Syndrome Disease Activity Index is a questionnaire that investigates the activity of SSP disease and has 12 domains (constitutional, lymphadenopathy, glandular, articular, cutaneous, respiratory, renal, muscular, peripheral nervous system, central nervous system, hematological, biological) (Seror et al. 2009). It was developed from a consensus study of the EULAR (European League Against Rheumatism) and the American group. His cross-cultural adaptation and validity for the Brazilian Portuguese language was performed by the Sjögren's syndrome clinic of the Rheumatology department of the Cassiano Antônio de Moraes University Hospital (HUCAM), in Vitória, Espírito Santo (Serrano et al., 2013). Disease activity is classified into 3 levels: mildly active, moderately active and highly active.

CONTACTS AND LOCATIONS:
Overall Officials: PAULO A MINALI, Principal Investigator — Federal University of São Paulo

IPD SHARING:
Plan to Share IPD: Yes
The questionaries SF-36 and ESSDAI used in the present study were shared with other researches.

REFERENCES:
- [Result] Baillet A, Vaillant M, Guinot M, Juvin R, Gaudin P. Efficacy of resistance exercises in rheumatoid arthritis: meta-analysis of randomized controlled trials. Rheumatology (Oxford). 2012 Mar;51(3):519-27. doi: 10.1093/rheumatology/ker330. Epub 2011 Nov 24. PMID 22120463
- [Result] Booth FW, Roberts CK, Laye MJ. Lack of exercise is a major cause of chronic diseases. Compr Physiol. 2012 Apr;2(2):1143-211. doi: 10.1002/cphy.c110025. PMID 23798298
- [Result] Cook DB, Nagelkirk PR, Poluri A, Mores J, Natelson BH. The influence of aerobic fitness and fibromyalgia on cardiorespiratory and perceptual responses to exercise in patients with chronic fatigue syndrome. Arthritis Rheum. 2006 Oct;54(10):3351-62. doi: 10.1002/art.22124. PMID 17009309
- [Result] O'Grady M, Fletcher J, Ortiz S. Therapeutic and physical fitness exercise prescription for older adults with joint disease: an evidence-based approach. Rheum Dis Clin North Am. 2000 Aug;26(3):617-46. doi: 10.1016/s0889-857x(05)70159-9. PMID 10989515
- [Result] Hakkinen A, Sokka T, Kautiainen H, Kotaniemi A, Hannonen P. Sustained maintenance of exercise induced muscle strength gains and normal bone mineral density in patients with early rheumatoid arthritis: a 5 year follow up. Ann Rheum Dis. 2004 Aug;63(8):910-6. doi: 10.1136/ard.2003.013003. PMID 15249317
- [Result] Peterson MD, Rhea MR, Sen A, Gordon PM. Resistance exercise for muscular strength in older adults: a meta-analysis. Ageing Res Rev. 2010 Jul;9(3):226-37. doi: 10.1016/j.arr.2010.03.004. Epub 2010 Apr 10. PMID 20385254
- [Result] Rooks DS, Silverman CB, Kantrowitz FG. The effects of progressive strength training and aerobic exercise on muscle strength and cardiovascular fitness in women with fibromyalgia: a pilot study. Arthritis Rheum. 2002 Feb;47(1):22-8. doi: 10.1002/art1.10180. PMID 11932874
- [Result] Stenstrom CH, Minor MA. Evidence for the benefit of aerobic and strengthening exercise in rheumatoid arthritis. Arthritis Rheum. 2003 Jun 15;49(3):428-34. doi: 10.1002/art.11051. No abstract available. PMID 12794800
- [Result] Champey J, Corruble E, Gottenberg JE, Buhl C, Meyer T, Caudmont C, Berge E, Pellet J, Hardy P, Mariette X. Quality of life and psychological status in patients with primary Sjogren's syndrome and sicca symptoms without autoimmune features. Arthritis Rheum. 2006 Jun 15;55(3):451-7. doi: 10.1002/art.21990. PMID 16739213
- [Result] Barendregt PJ, Visser MR, Smets EM, Tulen JH, van den Meiracker AH, Boomsma F, Markusse HM. Fatigue in primary Sjogren's syndrome. Ann Rheum Dis. 1998 May;57(5):291-5. doi: 10.1136/ard.57.5.291. PMID 9741313
- [Result] Belenguer R, Ramos-Casals M, Brito-Zeron P, del Pino J, Sentis J, Aguilo S, Font J. Influence of clinical and immunological parameters on the health-related quality of life of patients with primary Sjogren's syndrome. Clin Exp Rheumatol. 2005 May-Jun;23(3):351-6. PMID 15971423
- [Result] Dassouki T, Benatti FB, Pinto AJ, Roschel H, Lima FR, Augusto K, Pasoto S, Pereira RMR, Gualano B, de Sa Pinto AL. Objectively measured physical activity and its influence on physical capacity and clinical parameters in patients with primary Sjogren's syndrome. Lupus. 2017 Jun;26(7):690-697. doi: 10.1177/0961203316674819. Epub 2016 Oct 26. PMID 27798360
- [Result] d'Elia HF, Rehnberg E, Kvist G, Ericsson A, Konttinen Y, Mannerkorpi K. Fatigue and blood pressure in primary Sjogren's syndrome. Scand J Rheumatol. 2008 Jul-Aug;37(4):284-92. doi: 10.1080/03009740801907995. PMID 18612929
- [Result] Hackett KL, Newton JL, Frith J, Elliott C, Lendrem D, Foggo H, Edgar S, Mitchell S, Ng WF. Impaired functional status in primary Sjogren's syndrome. Arthritis Care Res (Hoboken). 2012 Nov;64(11):1760-4. doi: 10.1002/acr.21738. PMID 23111856
- [Result] Lendrem D, Mitchell S, McMeekin P, Bowman S, Price E, Pease CT, Emery P, Andrews J, Lanyon P, Hunter J, Gupta M, Bombardieri M, Sutcliffe N, Pitzalis C, McLaren J, Cooper A, Regan M, Giles I, Isenberg D, Vadivelu S, Coady D, Dasgupta B, McHugh N, Young-Min S, Moots R, Gendi N, Akil M, Griffiths B, Ng WF; UK primary Sjogren's Syndrome Registry. Health-related utility values of patients with primary Sjogren's syndrome and its predictors. Ann Rheum Dis. 2014 Jul;73(7):1362-8. doi: 10.1136/annrheumdis-2012-202863. Epub 2013 Jun 12. PMID 23761688
- [Derived] Minali PA, Pimentel C, de Mello MT, Lima G, Dardin LP, Garcia A, Goni T, Trevisani V. Effectiveness of resistance exercise in functional fitness in women with primary Sjogren's syndrome: randomized clinical trial. Scand J Rheumatol. 2020 Jan;49(1):47-56. doi: 10.1080/03009742.2019.1602880. Epub 2019 Jun 27. PMID 31244376